CLINICAL TRIAL: NCT05372471
Title: Efficacy of Using a Digital Platform for Diabetes Care Compared to Usual Care in Patients Diagnosed With Type 2 Diabetes Mellitus Type 2.
Brief Title: Efficacy of the Digital Platform for Diabetes Care Compared to Usual Care in Patients Diagnosed With Type 2 Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: FM-CIE-0689-19
Record Dates: First submitted 2022-05-08; First posted 2022-05-12 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Treated With Insulin
Keywords: Type 2 diabetes; Telemedicine; mHealth; ClouDi; Hospital
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Intervention Model Description: Randomized controlled clinical trial, not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mHealth (Other): Intervention group (mHealth platform users).
  Interventions: Other: mHealth
- Control (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: mHealth — ClouDi is a telemedicine platform that was developed for the remote monitoring of patients with diabetes in Colombia. It incorporated the recommendations that were published in a usability pilot study that was conducted previously with an open-source cloud platform. The platform consists of a web version, a version for mobile devices and a desktop application, which is installed on the patient's personal computer, thereby allowing glucose measurements taken through the Optium Neo glucometer (Abbott Diabetes Care, Alameda, CA, USA) to be uploaded automatically to the cloud. In this trial, the glucose measurements that were uploaded to the ClouDi website, were reviewed weekly by the members of the research group who were responsible for adjusting the therapy to the insulin titration scheme prescribed for the patient. The patients were informed about these adjustments by text messages sent from the web version of ClouDi to the patient's mobile phone via pop-up notifications.
  Arms: mHealth
Other: Usual Care — They will have a regular visit after 3 months where the capillary glucose data will be evaluated in person by the clinical team, the insulin dose will be titrated according to the type of insulin and the presence of hypoglycemia.
  Arms: Control

SUMMARY:
Introduction: In patients diagnosed with DM2, it is essential to achieve good metabolic control. One of the tools to optimize said control is self-monitoring with capillary glucometry or SMBG (Self Monitoring of Blood Glucose), which is indicated in all patients treated with insulin and is part of the "treat to target" strategies associated with education. Despite this, many patients do not perform self-titration of insulin due to the number of capillary glucose measurements (CG) necessary, or they do not record them adequately, which leads to therapeutic inertia. Digital platforms integrated with the use of smart mobile devices facilitate this process, and in experimental settings, they have shown a significant decrease in glycosylated hemoglobin (HbA1c) and an increase in adherence to therapy. However, at the moment there are no data about the efficacy of this system in the real population.

Objective: To determine the effectiveness of the use of a digital platform for diabetes care, in terms of HbA1c reduction, compared with the usual treatment, in patients with DM2 under follow-up in a chronic patient care center.

Methodology: A controlled clinical study will be carried out. Patients with a diagnosis of DM2, under follow-up in specialized centers, with poor glycemic control defined by HbA1c outside the goals and who have been discharged from a high complexity hospital will be included. Demographic, clinical, and insulin requirement variables will be recorded according to the total daily dose of insulin (DDT) in units. They will be randomly distributed into two groups; the intervention group will use SMBG integrated with a digital platform for diabetes care and the control group will use SMBG associated with usual care for 3 months. A comparison will be made between HbA1c levels, the number of episodes of severe hypoglycemia, nocturnal hypoglycemia, at baseline and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Poor metabolic control with HbA1C ≥ 8% and ≤ 11% measured using a method certified by the National Glycohemoglobin Standardization Program (NGSP), ≤ 3 months before the screening visit.
* Patients who use insulin therapy in the basal plus scheme, basal-bolus, or with two or more applications of insulin per day.
* Not having modified therapy in the last 3 months
* Availability of access to a computer to download data.
* Mobile access with data.
* The subject's compliance with capillary glucose self-monitoring parameters was greater than 80% during the baseline period after the Screening Visit.
* Accept the study including signing the informed consent

Exclusion Criteria:

* Acute decompensation of diabetes in the last 3 months
* History of myocardial infarction or acute coronary syndrome in the last three months before recruitment.
* Treatment with glucocorticoids in the last 3 months before the screening visit or who is scheduled to receive treatment during the study period
* Visual impairment that limits the ability to view or use the mobile application
* Cognitive impairment that, in the opinion of the principal investigator or study physician, would result in non-cooperation with study procedures.
* Active neoplastic disease or in the last year and/or life expectancy less than 6 months.
* Participating in another clinical study.
* Proliferative retinopathy, amputations attributable to diabetes, and/or severe peripheral neuropathy that could interfere with the ability to participate and follow the study.
* Pregnant or lactating, or plan to become pregnant during the study period
* Real-time or intermittent continuous glucose monitoring user.
* Significant psychiatric illness, kidney disease, severe liver disease, or other illness that affects the ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
HbA1c change | 3 months
  Evaluate the efficacy of a therapeutic strategy that integrates the use of a digital platform for diabetes care (CLOUDI) for 3 months, compared with usual care, in terms of HbA1c reduction, in patients with DM2 under follow-up in patient care centers chronic.

SECONDARY OUTCOMES:
Severe Hypoglycemia | 3 months
  To compare the incidence of severe hypoglycemia events in the 3 months of follow-up, in patients with DM2 users of the digital platform, and patients in usual management.
Hypoglycemia level 1 and 2 | 3 months
  To compare the incidence of global and nocturnal alert events (<70mg/dl) and clinically significant hypoglycemia (<54mg/dl) in patients with DM2.

CONTACTS AND LOCATIONS:
Overall Officials: Ana M Gómez Medina, Dr, Principal Investigator — Hospital Universitario San Ignacio
Locations (1):
- Hospital San Ignacio Hospital San Ignacio, Bogota, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make the iPad and related data available after we gain acceptance for the publishing article.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: Principal Investigator Approval